CLINICAL TRIAL: NCT05215223
Title: Effect of Whole Body Vibration on Insulin Resistance in Females With Polycystic Ovarian Syndrome
Acronym: WBV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Mohamed Ali Shehata, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003460
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Polycystic Ovarian Syndrome; Insulin Resistance
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance | interventions — Exercise Test

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- whole body vibration (Experimental): the patient will be received whole body vibration for three times/ week in addition to aerobic exercise for 3 times per week, 45 minutes per session for eight weeks
  Interventions: Device: whole body vibration; Device: Treadmill
- Aerboic exercise (Active Comparator): Moderate intensity aerobic exercise in form of walking on treadmill for 3 times per week, 45 minutes per session for eight weeks
  Interventions: Device: Treadmill

INTERVENTIONS:
Device: whole body vibration — the patients will stand on whole body vibration device with maintaining squatting position while keeping their trunk extended. The first training session will be consisted of three sets of 1 min and will be separated by a 1-min of standing rest. intensity will 1 mm. Then one set will be added every session
  Arms: whole body vibration
Device: Treadmill — Females will be asked to perform moderate intensity aerobic exercise for 45 minutes for 3 times per week for 8 weeks

SUMMARY:
The purpose of this study is to investigate the effect of whole body vibration on insulin resistance in females with polycystic ovarian syndrome

DETAILED DESCRIPTION:
polycystic ovarian syndrome is a complex endocrine condition characterized by metabolic abnormalities such as insulin resistance, excess weight or obesity, diabetes, and an increased risk of cardiovascular disease.Despite previous studies reported that physical exercise improves insulin resistance in females with polycystic ovarian syndrome, there is no study yet investigate the effect of whole body vibration on insulin resistance

ELIGIBILITY:
Inclusion Criteria:

1. Females with polycystic ovarian syndrome.
2. Their ages will range from 20 to 35 years.

Exclusion Criteria:

* 1-Smoking. 2-History of chronic disease.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 46 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Homeostasis Model Assessment (HOMA-IR) | eight weeks
  Estimate insulin resistance (IR), it will be calculated according to the formula: fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5.

SECONDARY OUTCOMES:
Waist circumference | eight weeks
  by a tape measurement around the waist
waist hip ratio | eight weeks
  The formula = waist circumference / hip circumference.
LH/FSH ratio | Eight weeks
  To assess the severity of PCOS

CONTACTS AND LOCATIONS:
Overall Officials: Mai M Ali Shehata, lecturer, Principal Investigator — faculty of physical therapy
Locations (1):
- Faculty of physical therapy, Giza, Egypt